CLINICAL TRIAL: NCT07064265
Title: Assessment of Interprofessional Competencies of Healthcare Professionals Before and After Healthcare Simulation Sessions
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0041_ECIPS
Record Dates: First submitted 2025-05-20; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-05

CONDITIONS: Health Personnel; Interprofessional Relations; CONTINUING MEDICAL EDUCATION

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to assess the interprofessional competencies of healthcare learners before and one month after interprofessional simulation sessions, and to demonstrate their impact on the work of healthcare professionals as part of their continuing education in a hospital setting.

Initially, we will distribute a self-assessment questionnaire to all learners before the simulation sessions and again one month after the sessions.

Hospital-based healthcare professionals register for the simulation training through the continuing education department of Gonesse Hospital.

Physicians and medical students register through the training's designated physician.

Paramedical students register through the training's designated nurse manager.

We conduct two simulation training sessions per month on the topic of "Adult Life-Threatening Emergencies: Cardiac Arrest."

Each session is composed of an interprofessional group.

Before the start of the session, the questionnaire is distributed to all participants.

Learners are asked to indicate only their profession and the date on the questionnaire.

Each questionnaire is assigned a number in the order of collection to ensure anonymity.

One month later, we resend the same questionnaire by email to the participants.

This is a self-assessment questionnaire developed in Canada and scientifically validated, used to evaluate interprofessional collaboration competencies (Survey for the Achievement of Interprofessional Collaborative Competencies: SACCI).

In a second phase, we will compare the results of the self-assessment questionnaires completed before and one month after the simulation sessions, using statistical analysis via Excel spreadsheet.

ELIGIBILITY:
Inclusion Criteria:

* Medical students (interns and externs)
* Paramedical students (nursing students, nurse assistants, nurse managers)
* Healthcare professionals from Gonesse Hospital

Exclusion Criteria:

* Administrative staff
* Participants who have already taken part in previous simulation sessions

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of healthcare learners and professionals involved in patient care and training at Gonesse Hospital (France). This includes medical students (interns and externs), paramedical students (such as nursing students, nurse assistants, and nurse managers), and hospital-based healthcare providers. Participants will be selected from those who voluntarily enroll in interprofessional simulation training sessions focused on adult life-threatening emergencies (cardiac arrest), as part of their continuing education or academic curriculum.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in interprofessional collaboration competencies of healthcare learners, as assessed by the SACCI questionnaire (Survey for the Achievement of Interprofessional Collaborative Competencies), between baseline (pre-simulation) and one month post-simul | May 2025 - March 2026

CONTACTS AND LOCATIONS:
Locations (1):
- France, Gonesse, France, France